CLINICAL TRIAL: NCT01194193
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of the m-Tor Kinase Inhibitor AZD8055 Using Intermittent Dosing Schedules in Patients With Advanced Solid Malignancies and Lymphomas
Brief Title: Preliminary Anti-tumour Activity of mTor Kinase Inhibitor in Advanced Tumours
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Amendment to study compound development programme
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1600C00002
Record Dates: First submitted 2010-08-18; First posted 2010-09-02 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Cancer; Advanced Solid Tumours; Lymphomas
Keywords: Cancer; Advanced solid tumours; lymphomas; dose escalation; preliminary anti-tumour activity; Tor kinase inhibitor; oral administration; intermittent dosing
MeSH Terms: conditions — Neoplasms; Lymphoma | interventions — (5-(2,4-bis((3S)-3-methylmorpholin-4-yl)pyrido(2,3-d)pyrimidin-7-yl)-2-methoxyphenyl)methanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AZD8055

INTERVENTIONS:
Drug: AZD8055 — Oral tablet, single dose on Day 1, followed by a 48 hour - 7 day washout and then either twice daily alternate days dosing from multiple dose day 1 onwards or twice daily dosing for 21 days from multiple dose day 1 onwards followed by 7 days no treatment. Cycles of 28 days.

SUMMARY:
To investigate the safety and tolerability of AZD8055 intermittent dosing schedules when given orally to patients with advanced solid malignancies and lymphomas. Two intermittent dosing schedules will be explored with increasing doses until a maximum tolerated dose is determined for each schedule.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological confirmation of an advanced solid malignant tumour or lymphoma which is refactory to standard therapies or for which no standard therapy exists, patients with measurable or non-measurable disease (according to RECIST criteria)
* WHO performance status 0-2
* Evidence of post-menopausal status or negative urine/serum pregnancy test for pre-menopausal female patients

Exclusion Criteria:

* Patients with severe laboratory abnormalities for haematology, liver or renal function. Also treatment with any haemopoietic growth factors are not allowed within two weeks from first dose of study drug.
* Any investigational agents or study drugs from a previous clinical study within 30 days, any other chemotherapy, immunotherapy or anticancer agents within 3 weeks of the first dose of study treatment
* Patients with severe cardiac condition of ischemia, impaired ventricular function and arrhythmias, evidence of severe or uncontrolled systemic or current unstable or uncompensated respiratory or cardiac conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 5), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 6), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 7), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 8), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 9), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 10), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 11), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 12), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 13), although safety and tolerability parameters will be measured at all visits.
Safety and tolerability of AZD8055; The number of patients with adverse events, including changes in vital signs, general organ function, clinical chemistry, haematology, urinalysis and physical examinations. | Evaluability period is 5 weeks (visit 14), although safety and tolerability parameters will be measured at all visits.
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 2)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 3)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 4)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 6)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 7)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 8)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 9)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 10)
Evaluate the pharmacokinetics of AZD8055; Pharmacokinetic analysis of the plasma and urine concentration data for AZD8055 and its metabolites will be performed following both single and multiple dosing with two intermittent dosing schedules. | 1 cycle (3-4 weeks, at visit 11)

SECONDARY OUTCOMES:
Preliminary assessment of the anti-tumour activity of AZD8055; Evalution of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1 and percentage change in tumour size and measurement of serological biomarkers. | Every 2 cycles (at visits 1, 17, every subsequent 8 weeks, visit 100
Investigation of possible relationships between plasma AZD8055 concentrations / exposure and changes in safety parameters (including number and types of adverse events). | 1 cycle (3-4 weeks, at visits 2, 3, 4, 6-11)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, MD, Study Director — AstraZeneca R&D